CLINICAL TRIAL: NCT00340951
Title: Can Immune Parameters Predict Acute and Chronic Rejection in Lung Recipients?
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905183; 05-E-N183
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-04-13

CONDITIONS: Lung Transplantation
Keywords: Regulatory T Cells; Bronchiolitis Obliterans Syndrome; Genetic Polymorphism; Innate Immunity; Transplantation; Lung Transplantation
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

SUMMARY:
This study will evaluate the ability of lung transplant recipients to react to the transplanted organs. Previous research indicates that some immune tests can identify whether people are at risk for chronic rejection of transplanted lungs. Certain parameters, that is, physical properties involving the immune system, may cause acute chronic rejection of the lungs, which may lead to chronic rejection, a condition of scarring that worsens lung function. If such parameters can be identified and distinguished from those found in healthy subjects, information gained can help medical professionals to provide individualized treatments that work on the immune system. Short-term and long-term survival of lung transplant recipients may thus be improved.

Patients who will have or have had lung transplants will be recruited by clinical transplant coordinators. Normal control subjects will be recruited through flyers and newspaper advertisements.

Collection of blood samples will be done at Duke University Medical Center. Blood collections will be done of patients undergoing routine pretransplant and posttransplant blood tests, so no extra blood collections will be required. Control subjects will undergo three blood collections over an 8-week period. They will be compensated for their time in participating, at the rate of $5 for the initial blood draw, $10 for the second one, and $15 for the third one. A small amount of blood is involved, about 3 tablespoons. The blood cells and DNA (which contains genetic material) will be isolated for analysis. Patients' DNA samples collected will be identified by a code, and all other identifying information will be removed. The samples may be used in the future as new tests are developed.

This study will not have a direct benefit for participants. However, during the study, if it is found that any patients have an inherited risk for a disease likely to cause early death if the disease is not treated, then the researchers will attempt to notify those patients. Overall, it is hoped that information gathered will enhance researchers' understanding of what tests best identify patients at risk for developing chronic rejection of their transplanted lungs.

DETAILED DESCRIPTION:
The aim of this study is to provide insight into the immune mechanisms involved in the pre- and posttransplant response of lung recipients to determine if short- and long-term graft outcome can be predicted and to allow for potential intervention. We have assembled a panel of assays that will test various functions of the immune response and investigate immune mechanisms involved in acute and chronic rejection (CR). Our overall hypothesis is that measurment of pre- and posttransplant immune response to donor HLA antigens/peptides can predict graft outcome. Our goal is to determine if immune parameters [ELISpot], intracellular T regulatory cells and ATP synthesis can identify lung recipients at high risk for developing AR and sub-clinical rejection. Sub-aim: To determine the correlation of cytokine genotypes with ELISpot results and T regulatory cell level and activity for recipients at high risk for developing acute rejection in comparison to a normal subject cohort. A second hypothesis is that recipients who experience an AR episode and remain responsive to donor antigen and those who show increased reactivity to donor HLA peptides are at high risk for developing CR. Our goal is to determine if the immune parameters (CFSE responder frequencies and response to donor peptides are assayed by CFSE, ELISpot, T regulatory cell level, and ATP synthesis) can identify lung recipients at high risk for developing CR and distinguish these immune parameters from a normal subject cohort. If successful, we will provide clinicians with the information necessary for individualization of immunosuppression intervention aimed at improving short and long-term graft outcome.

ELIGIBILITY:
* INCLUSION/EXCLUSION CRITERIA:

Adult patients undergoing transplant at Duke Medical Center are to be recruited as subjects.

In addition, investigators will recruit 80 adult control subjects from individuals who will not have lung disease and will not be on immunosuppression or from pre transplant subjects.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2005-06-23; Study Completion 2007-04-13

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - NIEHS, Research Triangle Park, Research Triangle Park, North Carolina